CLINICAL TRIAL: NCT00899288
Title: Investigating the Chemical Properties of Fingernails to Determine the Efficacy of Nail Structure for Evaluating Bone Fragility
Brief Title: Fingernails in Evaluating Bone Health in Postmenopausal Women With Breast Cancer Undergoing Hormone Therapy on Clinical Trial IBCSG-1-98
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Insufficient accrual
Sponsor: ETOP IBCSG Partners Foundation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CDR0000482403; IBCSG-18-98-FPS (Other: International Breast Cancer Study Group); IBCSG-1-98-FPS (Other: International Breast Cancer Study Group); EU-20625
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2012-07-27 (Estimated); Status verified 2012-07

CONDITIONS: Breast Cancer; Osteoporosis
Keywords: osteoporosis; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms; Osteoporosis | interventions — Spectrum Analysis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- tamoxifen and no bone fracture (Experimental): Patients randomized to Arm A of Study BIG 1-98 (tamoxifen for 5 years) who have not had a bone fracture.
  Interventions: Procedure: spectroscopy
- Letrozole and no bone fracture (Experimental): Patients randomized to Arm B of Study BIG 1-98 (letrozole for 5 years) who have not had a bone fracture.
  Interventions: Procedure: spectroscopy
- Tamoxifen and bone fracture (Experimental): Patients randomized to Arm A of Study BIG 1-98 (tamoxifen for 5 years) who have had a bone fracture.
  Interventions: Procedure: spectroscopy
- Letrozole and bone fracture (Experimental): Patients randomized to Arm B of Study BIG 1-98 (letrozole for 5 years) who have had a bone fracture.
  Interventions: Procedure: spectroscopy

INTERVENTIONS:
Procedure: spectroscopy — Nails will be chemically characterized using Raman spectroscopy.

SUMMARY:
RATIONALE: Studying samples of fingernails in the laboratory from patients with breast cancer may help in evaluating bone health in postmenopausal women undergoing hormone therapy for breast cancer.

PURPOSE: This laboratory study is examining fingernails as a way of evaluating bone health in postmenopausal women with breast cancer undergoing hormone therapy on clinical trial IBCSG-1-98.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the effects of tamoxifen vs letrozole on the chemical properties of fingernails by Raman spectroscopy in postmenopausal women with breast cancer undergoing adjuvant hormonal therapy on protocol IBCSG-1-98.
* Determine the efficacy of nail structure for evaluating bone fragility.

Secondary

* Compare fingernail assessments in patients who have had a bone fracture vs those who have not.
* Determine the natural variation in chemical (Raman spectroscopy) properties of 2 fingernails sourced at 1 appointment from the same donor.
* Evaluate the effect of further drug treatment (after 6 months) on the chemical properties of fingernails.

OUTLINE: This is a single-blind, multicenter, pilot study. Patients are stratified according to treatment on protocol IBCSG-1-98 (tamoxifen vs letrozole) and bone fracture (yes vs no).

Fingernail clippings are collected at baseline and 6 months later. Fingernail clippings are examined by Raman spectroscopy.

PROJECTED ACCRUAL: A total of 60 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Enrolled on protocol IBCSG-1-98

  * Currently receiving (i.e., have not yet completed) 5 years of treatment with tamoxifen or letrozole and expected to receive ≥ 6 months of additional treatment on protocol IBCSG-1-98
* No recurrent breast cancer or second primary cancer
* No known bone disease (including osteomalacia or osteogenesis imperfecta)
* Hormone receptor status

  * Estrogen and/or progesterone receptor positive tumor

PATIENT CHARACTERISTICS:

* Female
* Postmenopausal
* No uncontrolled thyroid or parathyroid disease, Cushing's disease, or other pituitary diseases
* No malabsorption syndrome or clinically relevant vitamin D deficiency

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 1 year since prior and no concurrent anticonvulsants
* More than 6 months since prior and no concurrent corticosteroids at doses > the equivalent of 5 mg/day of prednisone for > 2 weeks total
* No prior or concurrent sodium fluoride at daily doses ≥ 5 mg/day for > 1 month
* More than 12 months since prior and no concurrent anabolic steroids
* More than 6 months since any prior drug for the prevention of osteoporosis (excluding calcium or cholecalciferol [vitamin D])
* Concurrent warfarin allowed provided duration of treatment is no more than 4 weeks

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2005-04; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Determination of bone health using fingernail assessments at baseline and 6 months | At baseline and 6 months after inclusion in the trial

CONTACTS AND LOCATIONS:
Overall Officials: Mark Towler, MD, Study Chair — Materials & Surface Science Institute at the University of Limerick